CLINICAL TRIAL: NCT06847828
Title: The Effectiveness of Using a Palliative Care Question Prompt List on the Selfefficacy and Preparedness of Indonesian Homecare Workers in Providing End-of-Life Care to Terminally Ill Patients
Brief Title: The Effectiveness of Using a Palliative Care QPL on the Selfefficacy and Preparedness of Indonesian Homecare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Den,Yu-Yun (Other)
Responsible Party: Sponsor-Investigator, Den,Yu-Yun, student, Tzu Chi University
Organization: Tzu Chi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB112-186-B
Record Dates: First submitted 2025-01-23; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Question Prompt List; Caregivers; End-of-life Care

STUDY DESIGN:
Intervention Model Description: randomized control-group pretest-posttest design
Who Masked: Participant
Masking Description: single-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): During recruitment, the researcher contacts participants 1-3 days before the nurse's visit to explain the study and obtain consent. After signing, participants complete a pretest questionnaire and are randomly assigned to the experimental or control group.
  To assess baseline question-asking ability, the researcher first asks if participants have any caregiving-related questions. The intervention group receives the Indonesian QPL, consent form, and questionnaire, with instructions on QPL use.
  Within three days post-pretest, the researcher observes a nurse's visit without interfering, recording participant questions with consent. After the health education session, posttest data on end-of-life care preparedness, communication self-efficacy, and satisfaction are collected.
  Interventions: Other: QPL
- control group. (No Intervention): During recruitment, the researcher contacts participants 1-3 days before the nurse's visit to explain the study and obtain consent. After signing, participants complete a pretest questionnaire and are randomly assigned to the experimental or control group.
  To assess baseline question-asking ability, the researcher first asks if participants have any caregiving-related questions. The control group receives an Indonesian consent form and questionnaire, with usual health education provided by nurses. Translation support is available if needed.
  Within three days post-pretest, the researcher observes a nurse's visit without interfering, recording participant questions with consent. Afterward, posttest data on end-of-life care preparedness, communication self-efficacy, and satisfaction are collected.

INTERVENTIONS:
Other: QPL — The QPL is in the form of a structured list of questions that caregivers would like to ask. It includes 17 questions on concept communication and 20 questions on end-of-life care. You can check the questions you want to ask and then discuss them with the medical team.
  Arms: Experimental Group

SUMMARY:
Foreign studies on caregivers' use of QPL in end-of-life care, decision-making, and satisfaction are mostly conducted with family members who share the same language. Foreign family caregivers are a local cultural feature of Taiwan. This study explores the role of foreign family caregivers in end-of-life care in Taiwan. Cultural issues and differences, whether the number of questions asked, care readiness and self-efficacy can be increased after the intervention of the end-of-life care QPL, and the use of QPL that is appropriate for Indonesian culture to communicate and prepare for end-of-life care in hospice home care, is expected to provide A reference for communication between medical teams and foreign home caregivers and improvement of care quality.

DETAILED DESCRIPTION:
Research Background and Purpose Since Taiwan allowed the employment of foreign family caregivers in 1992, the proportion of caregiving roles taken up by these workers has steadily increased. However, many foreign family caregivers lack the cognitive and social skills needed for end-of-life care. When faced with challenges, they often resort to sending patients back to the hospital, resulting in higher medical costs. These caregivers frequently do not know what to expect or how to ask relevant questions, underscoring the need for clear information to assist them in communicating with healthcare teams. The Question Prompt List (QPL) is a simple, personalized, and cost-effective tool that helps individuals structure their thoughts, ask questions, gain a sense of control, gather information, and facilitate communication between caregivers and healthcare providers.

Although there has been increasing domestic research on the caregiving abilities and stress of foreign caregivers, studies on communication tools for end-of-life care are limited. Internationally, research on the use of QPLs in end-of-life caregiving often focuses on family members sharing a common language, but Taiwan's reliance on foreign caregivers presents unique cultural characteristics. This study explores the challenges and cultural differences experienced by foreign caregivers in Taiwan's end-of-life care setting. It examines whether using a culturally appropriate QPL tailored to Indonesian caregivers can enhance the number and quality of questions raised during communication and improve the overall effectiveness of communication. The findings are expected to provide valuable insights for improving communication and care quality between healthcare teams and foreign caregivers. Research Method V This study adopts a two-group randomized experimental design supplemented by qualitative data analysis to evaluate the effectiveness of a QPL in end-of-life care. The participants are Indonesian caregivers working in hospice wards or providing home care at a medical center in eastern Taiwan. The experimental group received QPL intervention as part of end-of-life care education and communication, while the control group received standard education and communication guidance. The outcome measures include self-designed questionnaires assessing communication self-efficacy, caregiving preparedness, and communication satisfaction. Paired t-tests and ANCOVA were used to analyze differences between pretest and posttest results within and between groups. Qualitative data were collected through feedback records during the communication guidance process and semi- structured interviews to gather participants' experiences and perceptions of using the QPL.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are fluent in Mandarin or Indonesian and have no reading or hearing impairment;
2. Agree to accept the commission and the Taxation Committee issues a letter of approval for the legal Indonesian guardian

Exclusion Criteria:

1. Those who are unable to communicate in Mandarin or Indonesian;
2. The employer of the patient has changed jobs and the patient cannot be contacted after the patient passes away;
3. Those who are under great pressure of end-of-life care or are physically unfit to take the questionnaire

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
caregiving preparedness | 3 days
  The scale assesses two aspects: "Preparedness for Patient Care" and "Preparedness for Caregiving Situations." A score of 1 indicates no preparedness, while 10 indicates full preparedness. Higher scores reflect greater perceived readiness.
communication self-efficacy | 3days
  The communication self-efficacy measure was designed to measure the Indonesian home caregivers' ability and confidence in the communication process, with a total of 7 questions. Respondents responded on a scale of 1-10, with 1 being "very unconfident", 5 being "average", and 10 being "very confident".Higher scores reflect greater self-efficacy.
satisfaction levels | 3days
  Communication satisfaction questionnaire. The control group had 9 questions and the intervention group had 15 questions (including the experience of using the end-of-life care questionnaire). 1 is "not prepared at all", 2 is "somewhat prepared", 3 is "average", 4 is "mostly prepared", and 5 is "very prepared". The higher the score, the higher the satisfaction.
number of questions asked education communication | 3days
  Within 3 days after the pretest, the researcher and the nurse visited the case together. During the visit, the researcher was a bystander and did not intervene in the communication and interaction between the nurse and the case. He only recorded the case's questions during the interaction process and asked for consent during the interaction process. The results were recorded in the form of audio recordings. The experimental group asked an Indonesian home care worker to review the content, circle or ask questions they wanted to know. The results of the audio recordings of the research process were translated into text and analyzed by two senior nurses with a master's degree or above. After the analysis was completed, the researcher and the two analysts held a consensus meeting to communicate on the inconsistent parts. The completed result is to calculate the number of questions asked in the communication interaction process.

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Mei Chang, Study Director — Ph.D
Locations (1):
- Tzu Chi University, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No